CLINICAL TRIAL: NCT05738252
Title: Frailty Assessments for Risk Assessment in Gynecologic Oncology Patients Undergoing Surgery and Chemotherapy
Brief Title: Frailty Assessments for Risk Assessment in Gynecologic Oncology Patients
Acronym: FARGO
Status: Recruiting | Type: Observational
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: v1.0_20211130
Record Dates: First submitted 2023-01-31; First posted 2023-02-22 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Gynecologic Cancer; Frailty; Oncology
MeSH Terms: conditions — Frailty; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Only participants providing specific separate consent will be enrolled in the biobank study. We will collect blood samples from patients at baseline, i.e., before and after starting the NACT and/or before surgery, and then at 28 days after surgery, 6 months and 12 months. We will collect EDTA tubes to obtain both plasma and whole blood for DNA analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group A: We expect that some of the eligible patients (Group A) will undergo surgery without NACT. Group A will undergo only one preoperative study visit (baseline) within 45 days prior to their surgery. Group A will complete the study assessments and follow-ups. Some patients of Group A will undergo adjuvant chemotherapy after surgery; this will not affect their study timeline.
  Interventions: Diagnostic Test: Clinical Frailty Scale; Diagnostic Test: Frailty Phenotype
- Group B: Patients undergoing NACT before their surgery (group B) will have a first baseline study assessment within 45 days prior to their first chemotherapy treatment; in this group, a second preoperative study visit will be repeated after chemotherapy is considered terminated at least 18 days post-chemotherapy cycle and within 45 days prior to surgery. Group B will complete the study assessments and follow-ups. Some patients of Group B will undergo adjuvant chemotherapy after surgery; this will not affect their study timeline.
  Interventions: Diagnostic Test: Clinical Frailty Scale; Diagnostic Test: Frailty Phenotype
- Group C: Post-chemotherapy, a small proportion of patients will not be deemed eligible for surgery by the treating physician (group C). Group C will be included in the evaluation of chemotherapy-related outcomes, and will also be asked to complete a follow-up visit 6 months from the date of registration
  Interventions: Diagnostic Test: Clinical Frailty Scale; Diagnostic Test: Frailty Phenotype
- Group D: An even smaller proportion of patients will initially be deemed eligible, recruited, and will complete the baseline assessment; however, they will eventually not undergo neither surgery nor chemotherapy. For Group D, a follow-up visit at 6 months from the baseline visit will be completed.
  Interventions: Diagnostic Test: Clinical Frailty Scale; Diagnostic Test: Frailty Phenotype

INTERVENTIONS:
Diagnostic Test: Clinical Frailty Scale — A way to summarize the overall level of fitness or frailty of an older adult after they had been evaluated by an experienced clinician
  Other Names: CFS
Diagnostic Test: Frailty Phenotype — Defined by the presence of three from the following five clinical features: weakness, slow walking speed, unintentional weight loss, exhaustion, and low physical activity
  Other Names: FP

SUMMARY:
FARGO is a prospective cohort study that aims to determine the performance of preoperative frailty assessment based on the Frailty Phenotype (FP), compared to a perioperative cardiovascular risk assessment based on the combination of preoperative Revised Cardiac Risk Index (RCRI), age and occurrence of myocardial injury after noncardiac surgery (MINS), in predicting the composite of all-cause death or new disability at 6 months after surgery in patients aged 55 or older. Patients will have confirmed or suspected gynecologic cancer, undergoing cytoreductive or high-risk surgery with or without chemotherapy.

DETAILED DESCRIPTION:
Little is known about how to best predict postoperative outcomes, recovery from complications, and chemotherapy tolerance in an increasingly older and medically complex GO population. Measuring frailty may represent a comprehensive tool for risk prediction. The study 1) will help fill the current gap in knowledge; 2) will translate into clinical practice changes both locally, and when replicated in a larger multi-centre study, elsewhere in Canada and worldwide; and 3) will inform future studies on shared decision-making strategies and interventions.

By evaluating the role of frailty as a static or dynamic predictor of patient important outcomes, and by considering the complexity of these patients and also of their treatment trajectories, the study has the potential to fill those gaps and influence how care is delivered. By involving stakeholders in the evaluation of feasibility and acceptability of frailty assessment, this will inform a change in care that is sustainable, innovative, and patient-centred.

There have been substantial knowledge advancements about perioperative risk factors and the long-term impact of postoperative complications; however, oncology patients and patient-reported outcomes have been insufficiently studied. There is increased literature on frailty assessment in noncardiac surgery; however, studies that included GO patients are few and of low-quality. The study will overcome the limitations of the current knowledge and practice, and will potentially change healthcare delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Age must be 55 years or older at registration
2. Must meet any one of the following criteria:

   1. Have stage II-IV ovarian or endometrial cancer, undergoing cytoreductive surgery via laparotomy, with or without neoadjuvant chemotherapy (NACT)
   2. Have any stage endometrial, uterine or cervical cancer planned for laparotomy where laparoscopy is deemed unfeasible/high-risk due to comorbidities
   3. Are undergoing laparotomy for pelvic mass, highly suspicious for malignancy; or
   4. Are undergoing laparotomy for gynecologic malignancy recurrence.

Exclusion Criteria:

1. Unable to provide informed consent
2. Require urgent surgery within 24 hours of first consultation to the Gynecological Oncology team
3. Are undergoing neoadjuvant radiation therapy
4. Have a previously documented history of dementia
5. Have cognitive, language, vision, or hearing impairment that impacts ability to understand the directions for the completion of the study instruments
6. Are participating in a clinical trial investigating a new systemic therapy

Ages: 55 Years to 110 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: FARGO will recruit patients aged 55 or older, with confirmed or suspected gynecologic cancer, undergoing cytoreductive or high-risk surgery with or without chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
All-cause death or new disability at 6 months | 6 months
  Disability status is determined using the 12-item World Health Organization Disability Assessment Schedule (WHODAS 2.0). New disability at any time point is based according to the following criteria that account for baseline disability scores:
  1. For individuals with a disability score of <25% at baseline, new disability is defined as a disability score ≥25% at follow-up;
  2. For individuals with a disability score ≥25%, new disability is defined an increase in disability score of ≥8%.
  Vascular death is defined as any death with a vascular cause and includes those deaths following a myocardial infarction, cardiac arrest, stroke, cardiac revascularization procedure (i.e., percutaneous coronary intervention [PCI] or coronary artery bypass graft [CABG] surgery), pulmonary embolus, hemorrhage, or deaths due to an unknown cause. Non-vascular death is defined as any death due to a clearly documented non-vascular cause (e.g. trauma, infection, malignancy).

SECONDARY OUTCOMES:
All cause death | 28 days and 1 year
  Vascular death is defined as any death with a vascular cause and includes those deaths following a myocardial infarction, cardiac arrest, stroke, cardiac revascularization procedure (i.e., percutaneous coronary intervention [PCI] or coronary artery bypass graft [CABG] surgery), pulmonary embolus, hemorrhage, or deaths due to an unknown cause. Non-vascular death is defined as any death due to a clearly documented non-vascular cause (e.g., trauma, infection, malignancy).
Oncologic Outcomes: Progression Free Survival (PFS) | at 6 and 12 months
  PFS, defined as the time from treatment initiation to tumor progression or recurrence or death from any cause, or to the date of censoring at the last time the subject was known to be alive. Cancer progression/recurrence will be defined as a measurable progression/recurrence documented on imaging.
Oncologic Outcomes: Cancer-specific death | at 6 and 12 months
  Cancer-specific death is death directly attributable to the primary gynecological cancer or directly related to its treatment, in the absence of other causes of death.
New Disability | 28 days, 6 months and 1 year after surgery
  Disability status is determined using the 12-item World Health Organization Disability Assessment Schedule (WHODAS 2.0). New disability at any time point is based according to the following criteria that account for baseline disability scores:
  1. For individuals with a disability score of <25% at baseline, new disability is defined as a disability score ≥25% at follow-up;
  2. For individuals with a disability score ≥25%, new disability is defined an increase in disability score of ≥8%.
  Definition of new disability at 28 days, 6 months, and 1 year after surgery will use as baseline disability score the WHODAS 2.0 score measured before surgery.
Major vascular complications | at 28 days, 6 months, and 1 year after surgery
  defined as a composite of vascular death, and non-fatal myocardial infarction (or myocardial injury for the 28-day time point), stroke, symptomatic proximal venous thromboembolism, and cardiac arrest
Infection, and infection with sepsis | at 28 days, 6 months, and 1 year after surgery
  Infection is defined as a pathologic process caused by the invasion of normally sterile tissue or fluid or body cavity by pathogenic or potentially pathogenic organisms.
  The Third International Consensus Definitions Task Force defines sepsis as a "life-threatening organ dysfunction due to a dysregulated host response to infection." Based on the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3) criteria, sepsis will require a quick Sequential Organ Failure Assessment (qSOFA) Score ≥2 points due to infection. The qSOFA includes the following items and scoring system:
  1. Altered mental status (1 point)
  2. systolic blood pressure of 100 mm Hg or less (1 point), and
  3. respiratory rate of 22 breaths/min or more (1 point).
In-hospital delirium | During the index hospital admission for surgery up to the first 3 days after surgery or before discharge from hospital
  Delirium during the first 3 days after surgery or before discharge from the hospital, based on Confusion Assessment Method (CAM). According to CAM, patients are diagnosed with delirium if they meet the first 2 criteria (acute onset with fluctuating course, AND attention deficit), and at least one of the second 2 criteria (disorganized thinking OR altered level of consciousness). Participants will be screened for postoperative delirium while in hospital, twice daily, during the first 3 days after surgery or until discharge (if before 3 days), by research personnel, using the 3D-CAM, or the CAM-ICU any time the participants are in the PACU or in ICU
Bleeding Independently Associated with Mortality after noncardiac Surgery | 28 days after surgery
  BIMS is a bleeding meeting any of the following 3 criteria:
  1. Leading to a postoperative hemoglobin <70 g/L
  2. Requiring transfusion of one or more units of red blood cells
  3. Judged to be the immediate cause of death
Acute congestive heart failure | 28 days after surgery, 6 months and 1 year after surgery
  The definition of congestive heart failure requires at least one of the following clinical signs (i.e. any of the following signs: elevated jugular venous pressure, respiratory rales/crackles, crepitations, or presence of S3) and at least one of the following:
  1. Radiographic findings (i.e., vascular redistribution, interstitial pulmonary edema, or frank alveolar pulmonary edema) OR
  2. Heart failure treatment implemented with diuretics with documented clinical improvement.
Unplanned admission to ICU | during index hospitalization for surgery
  admission to the ICU that was not planned
New clinically important atrial fibrillation | 28 days after surgery, 6 months and 1 year after surgery
  The definition of new clinically important atrial fibrillation requires the documentation of atrial fibrillation or atrial flutter of any duration on an ECG or rhythm strip, which results in angina congestive heart failure, symptomatic hypotension, or requires treatment with a rate controlling drug, antiarrhythmic drug, or electrical cardioversion.
Length of stay | during index hospitalization for surgery
  time spent in hospital immediately after surgery
Chemotherapy-related outcomes: total dose received | Before Surgery, 6-months post-surgery
  This will be measured at the end of any chemotherapy treatment when considered terminated:
  Total dose received, defined as Relative Dose Intensity (RDI), as calculated as the percentage of the standard dose that was administered
Chemotherapy-related outcomes: time to completion of all chemotherapy cycles | Before Surgery, 6-months post-surgery
  This will be measured at the end of any chemotherapy treatment when considered terminated:
  Time to completion of all chemotherapy cycles (number of days)
Chemotherapy-related outcomes: patient's decisional regret | Before Surgery, 6-months post-surgery
  This will be measured at the end of any chemotherapy treatment when considered terminated:
  Patient's decisional regret, defined as "distress or remorse after a (health care) decision," assessed using the Decisional Regret scale, a validated a 5-item scale
Chemotherapy-related outcomes: Change in health-related function or well-being | Before Surgery, 6-months post-surgery
  This will be measured at the end of any chemotherapy treatment when considered terminated:
  Change in health-related function or well-being, defined as the difference in WHODAS 2.0 score after chemotherapy compared to before chemotherapy.
Chemotherapy-related outcomes | Before Surgery, 6-months post-surgery
  This will be measured at the end of any chemotherapy treatment when considered terminated:
  Change in health-related quality of life, defined as the difference in FACT-G7 score after chemotherapy compared to before chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Maura Marcucci, MD, Principal Investigator — Population Health Research Institute
Locations (4):
- Canada (4):
  - Juravinksi Hospital, Hamilton, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Sunnybrook, Toronto, Ontario
  - University Health Network, Toronto, Ontario

REFERENCES:
- [Derived] Nguyen JMV, Vicus D, Hogen L, Zigras T, Pare G, Chong M, Benitez YR, Devereaux PJ, Ofori S, Borges FK, Di Sante E, Miletic D, Panus O, Vincent J, Ramasundarahettige C, Nene S, Patel A, Marcucci M. Frailty Assessment for Risk prediction in Gynecologic Oncology patients undergoing surgery and chemotherapy (FARGO) study protocol: Rationale and design of a multi-centre prospective cohort study. PLoS One. 2025 Jul 28;20(7):e0325651. doi: 10.1371/journal.pone.0325651. eCollection 2025. PMID 40720507